CLINICAL TRIAL: NCT00077142
Title: Phase I/II Dose Escalation, Pharmacokinetic, Safety, and Efficacy Study of Oral TAC-101 in Patients With Advanced Hepatocellular Carcinoma
Brief Title: TAC-101 in Treating Patients With Advanced Hepatocellular Carcinoma (Liver Cancer)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-007; P30CA016672 (NIH); MDA-ID-01007 (Other: UT MD Anderson Cancer Center); TAIHO-TAC101; NCI-1528; CDR0000349508 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Liver Cancer
Keywords: advanced adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; Oral TAC-101
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — TAC 101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAC-101 (Experimental): Oral TAC-101 daily Days 1-14, repeats every 21 days for 2 courses.
  Interventions: Drug: TAC-101

INTERVENTIONS:
Drug: TAC-101 — Once daily by mouth on days 1-14, repeat every 21 days for 2 courses.

SUMMARY:
RATIONALE: TAC-101 may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: This phase I/II trial is studying the side effects and best dose of TAC-101 and to see how well it works in treating patients with advanced hepatocellular carcinoma (liver cancer).

DETAILED DESCRIPTION:
OBJECTIVES:

Phase I

* Primary

  * Determine the maximum tolerated dose (MTD) of TAC-101 in patients with advanced hepatocellular carcinoma.
  * Determine the safety of 2 consecutive courses of this drug in these patients.
  * Determine the pharmacokinetics of this drug in these patients.
  * Determine the toxic and adverse effects profile of this drug in these patients.

Phase II

* Primary

  * Determine the objective antitumor response rate in patients treated with this drug at the MTD.
* Secondary

  * Determine the overall survival time of patients treated with this drug.
  * Determine the time to disease progression in patients treated with this drug.
  * Determine the duration of observed objective response, using WHO criteria and measurements of serum alpha-fetoprotein concentrations, in patients treated with this drug.
  * Determine the time to treatment failure in patients treated with this drug.
  * Determine the safety and tolerability of intermittent treatment with this drug in these patients.

OUTLINE: This is an open-label, dose-escalation study.

* Phase I: Patients receive oral TAC-101 once daily on days 1-14. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of TAC-101 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive oral TAC-101 at the MTD (determined in phase I) once daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 35-60 days.

PROJECTED ACCRUAL: A total of 6-18 patients for the phase I portion and 21-41 patients for the phase II portion will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatocellular carcinoma
* At least 1 previously unirradiated, bidimensionally measurable lesion greater than 20 mm by MRI or conventional CT scan OR at least 10 mm by spiral CT scan
* Patients with CNS involvement must have completed appropriate treatment and have no progressive neurologic deficits within the past 28 days
* No carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* ECOG 0-2

Life expectancy

* More than 12 weeks

Hematopoietic

* Hemoglobin ≥ 10.0 g/dL
* WBC ≥ 2,000/mm^3
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 40,000/mm^3
* No abnormal bleeding or clotting

Hepatic

* No grade C Child-Pugh cirrhosis
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Albumin ≥ 2.8 g/dL
* INR ≤ 1.5 times ULN
* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No prior deep vein thrombosis
* No prior superficial venous thrombosis
* No family history of thromboembolism in a first-degree relative
* No lower extremity thromboses by Doppler ultrasound (unless a subsequent venous angiography confirms a false positive ultrasound)

Pulmonary

* No prior pulmonary embolism

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception, except oral contraceptives containing estrogen
* Fasting triglycerides ≤ 400 mg/dL for men or ≤ 325 mg/dL for women
* No other malignancy within the past 3 years except inactive nonmelanoma skin cancer or carcinoma in situ of the cervix
* No uncontrolled metabolic disorders, other nonmalignant organ or systemic disease, or secondary effects of cancer that induce a high medical risk
* No known allergy or hypersensitivity to TAC-101 or its components

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior thalidomide
* No prior putative antiangiogenesis therapy
* Prior interferon allowed

Chemotherapy

* No more than 2 prior chemotherapy regimens

Endocrine therapy

* No concurrent estrogen products

Radiotherapy

* See Disease Characteristics
* More than 21 days since prior radiotherapy, except small portal radiotherapy used for the palliation of isolated, symptomatic, osseous metastases
* No prior radiotherapy to evaluable lesions
* No concurrent radiotherapy unless for bone pain that is present before beginning study

Surgery

* Not specified

Other

* Prior anticancer treatment allowed provided there is clear evidence of progressive disease after the most recent treatment
* More than 21 days since prior anticancer therapy and recovered
* No more than 2 prior treatment regimens
* No concurrent therapeutic anticoagulants

  * Concurrent low-dose warfarin for prophylactic care of indwelling venous access devices allowed
* No concurrent azoles or tetracyclines
* No concurrent medications known or suspected to increase risk of venous thromboembolism
* No other concurrent retinoids

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2001-04; Primary Completion 2005-07 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of TAC-101 | 60 Days

CONTACTS AND LOCATIONS:
Overall Officials: Melanie B. Thomas, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- [Result] Higginbotham KB, Lozano R, Brown T, Patt YZ, Arima T, Abbruzzese JL, Thomas MB. A phase I/II trial of TAC-101, an oral synthetic retinoid, in patients with advanced hepatocellular carcinoma. J Cancer Res Clin Oncol. 2008 Dec;134(12):1325-35. doi: 10.1007/s00432-008-0406-2. Epub 2008 May 27. PMID 18504614
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org